CLINICAL TRIAL: NCT05352828
Title: Phase 1b Study Evaluating the Safety and Efficacy of Autologous CD30.CAR-T in Combination With PD-1 Checkpoint Inhibitor (Nivolumab) in Relapsed or Refractory Classical Hodgkin Lymphoma Patients After Failure of Frontline Therapy (ACTION)
Brief Title: Autologous CD30.CAR-T in Combination With Nivolumab in cHL Patients After Failure of Frontline Therapy
Acronym: ACTION
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tessa Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TESSCAR003
Record Dates: First submitted 2022-04-08; First posted 2022-04-29 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Classical Hodgkin Lymphoma; Hodgkin Disease Refractory; Hodgkin Disease Recurrent
Keywords: cHL
MeSH Terms: interventions — Nivolumab; fludarabine; fludarabine phosphate; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Upon successful leukapheresis to produce CD30.CAR-T cells, patients will enter the treatment phase of the study. Treatments will include 4 cycles of nivolumab and CD30.CAR-T infusion (preceded by lymphodepletion chemotherapy). Patients will then enter the post-treatment follow-up phase of the study, whereby patients will undergo either autologous stem cell transplant or continue to receive up to 6 additional treatment cycles of nivolumab. Patients will be followed for response assessments and safety monitoring until end of study (EOS); approximately 3 years after leukapheresis. Long-term follow-up will continue with additional safety monitoring and survival for up to 15 years after Leukapheresis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and CD30.CAR-T (Experimental): Study treatment will include 4 cycles of nivolumab and a single CD30.CAR-T infusion (preceded by lymphodepletion chemotherapy of Fludarabine and Bendamustine).
  Interventions: Drug: Nivolumab; Drug: Autologous CD30.CAR-T; Drug: Fludarabine; Drug: Bendamustine

INTERVENTIONS:
Drug: Nivolumab — Dose: 480 mg or 6 mg/kg Q4W
  Other Names: Opdivo
Drug: Autologous CD30.CAR-T — Dose: 2 x 10e8 cells/m2
  Other Names: CD30-directed CAR-T cells
Drug: Fludarabine — Dose: 30 mg/m2/day x 3 days
  Other Names: Fludara
Drug: Bendamustine — Dose: 70 mg/m2/day x 3 days
  Other Names: Bendeka; Treanda

SUMMARY:
This is a Phase 1b, multicenter, open-label, single arm study to evaluate the safety and efficacy of the combination therapy, CD30.CAR-T and the programmed cell death protein-1 (PD-1) checkpoint inhibitor, nivolumab, in patients aged 12 years of age and above with relapsed or refractory classical Hodgkin lymphoma (cHL) following failure of standard frontline therapy.

DETAILED DESCRIPTION:
Upon successful leukapheresis to produce CD30.CAR-T cells, patients will enter the treatment phase of the study. Treatments will include 4 cycles of nivolumab and CD30.CAR-T infusion (preceded by lymphodepletion chemotherapy). Patients will then enter the post-treatment follow-up phase of the study, whereby patients will undergo either autologous stem cell transplant or continue to receive up to 6 additional treatment cycles of nivolumab. Patients will be followed for response assessments and safety monitoring until end of study (EOS); approximately 3 years after leukapheresis. Long-term follow-up will continue with additional safety monitoring and survival for up to 15 years after Leukapheresis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF
2. Male or female patients who are 12 years of age and above
3. Relapsed or refractory CD30+ cHL following failure of a standard frontline chemotherapy
4. At least 1 lesion, which must be fluordeoxyglucose positron emission tomography (FDG-PET) avid and measurable by PET-CT scan
5. Adequate laboratory parameters including hematologic, renal, hepatic, and coagulation function
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, or equivalent either Karnofsky performance status (for patients ≥ 16 years of age) or Lansky performance status (for patients < 16 years of age)
7. Anticipated life expectancy > 12 weeks
8. No active infections including COVID 19 at Screening

Exclusion Criteria:

1. Evidence of lymphomatous involvement of the central nervous system (CNS)
2. Presence of clinically relevant or active seizure disorder, stroke, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with central nervous system (CNS) involvement
3. Symptomatic cardiovascular disease: Class III or IV according to the New York Heart Association (NYHA) Functional Classification
4. Active uncontrolled bleeding or a known bleeding diathesis
5. Inadequate pulmonary function defined as oxygen saturation by pulse oximetry < 90% on room air
6. Echocardiogram (ECHO) or Multi-gated Acquisition (MUGA) scan with left ventricular ejection fraction (LVEF) < 45%
7. Prior receipt of salvage therapy, for relapsed or refractory cHL, including allogeneic or ASCT
8. Prior receipt of investigational CD30.CAR-T cells
9. Receiving any investigational agents or any tumor vaccines
10. Receiving any live/attenuated vaccines
11. Ongoing treatment with immunosuppressive drugs or chronic systemic corticosteroids
12. Unresolved > Grade 1 non-hematologic toxicity associated with any prior treatments
13. Previous history of known or suspected autoimmune disease within the past 5 years
14. Active interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
15. Evidence of human immunodeficiency virus (HIV) infection
16. Evidence of active viral infection with hepatitis B virus (HBV)
17. Evidence of active viral infection with hepatitis C virus (HCV)
18. Active second malignancy or history of another malignancy within the last 3 years
19. History of hypersensitivity reactions to murine protein-containing products or other product excipients
20. Any allergic or adverse reaction to nivolumab, fludarabine, or bendamustine that precludes treatment with these agents
21. History of a significant irAE from prior immune checkpoint inhibitor therapy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2037-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety of autologous CD30.CAR-T in combination with nivolumab | From first dose of nivolumab (Cycle 1) to end of nivolumab Cycle 4 (each cycle is 28 days)
  DLT

SECONDARY OUTCOMES:
Anti-tumor activity using CR rate of autologous CD30.CAR-T in combination with nivolumab | Up to end of 10 weeks post-CD30.CAR-T treatment
  CR rate
Overall response rate | Through study completion, an average of 3 years from Leukapheresis
  ORR
Duration of response | Through study completion, an average of 3 years from Leukapheresis
  DOR
Progression-free survival | Through study completion, an average of 3 years from Leukapheresis
  PFS

OTHER OUTCOMES:
Overall survival | Through study completion, an average of 3 years from Leukapheresis
  OS
Pharmacokinetics - Maximum concentration (Cmax) | Through study completion, an average of 3 years from Leukapheresis
  Maximum concentration of CD30.CAR-T
Pharmacokinetics - Time of maximum concentration (Tmax) | Through study completion, an average of 3 years from Leukapheresis
  Time to peak concentration of CD30.CAR-T in the blood
Pharmacokinetics - Area under the curve | Through study completion, an average of 3 years from Leukapheresis
  Area under the curve of CD30.CAR-T in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine; Sairah Ahmed, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - University of Miami, Miami, Florida
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No